CLINICAL TRIAL: NCT06392295
Title: A Phase II Trial of PSMA-Directed Para-Aortic Radiation Therapy for Oligorecurrent Prostate Cancer - The OCEAN Trial
Brief Title: PSMA-Directed Para-Aortic Radiation Therapy for Oligorecurrent Prostate Cancer
Acronym: OCEAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Benjamin Rich, Assistant Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231278
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Hormone Sensitive Prostate Cancer
Keywords: Oligorecurrent Disease
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PSMA-Guided PA-RT Group (Experimental): Participants in this group will undergo up to six months of systemic androgen deprivation therapy (ADT) and Androgen receptor signaling inhibitor (ARSI). During system therapy, participants will undergo five weeks of para-aortic radiation therapy.
  Total participation duration is up to five years.
  Interventions: Radiation: Para Aortic Radiation Therapy: Photon Therapy; Radiation: Para Aortic Radiation Therapy: Proton Therapy; Drug: Androgen Deprivation Therapy; Drug: Androgen Receptor Signaling Inhibitor

INTERVENTIONS:
Radiation: Para Aortic Radiation Therapy: Photon Therapy — Participants will undergo five weeks of PA-RT daily, for up to 30 minutes per day for 25 days, Monday through Friday, consisting of a total dose of 50 grays (Gys) delivered in 25 fractions to the Clinical Tumor Volume (CTV).
  Other Names: PA-RT Photon Therapy
Radiation: Para Aortic Radiation Therapy: Proton Therapy — Participants will undergo five weeks of PA-RT daily, for up to 30 minutes per day for 25 days, Monday through Friday, consisting of a total dose of 60 to 65 Gys delivered in 25 fractions to the Gross Tumor Volume (GTVn).
  Other Names: PA-RT Proton Therapy
Drug: Androgen Deprivation Therapy — Androgen deprivation therapy will be administered as per standard of care.
  Other Names: ADT
Drug: Androgen Receptor Signaling Inhibitor — Androgen receptor signaling inhibitor (ARSI) will be administered as per standard of care.
  Other Names: ARSI

SUMMARY:
The purpose of this prostate cancer research study is to learn about:

1. Improving control of prostate cancer using radiation therapy, delivered to the para-aortic and pelvic lymph nodes, in addition to systemic androgen suppression therapy;
2. Preserving quality of life after radiation therapy;
3. Leveraging imaging results from prostate-specific membrane antigen (PSMA) positron emission tomography (PET)/computed tomography (CT) scans to evaluate and manage disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven prostate adenocarcinoma
2. Male, ≥ 18 years old
3. Oligorecurrent disease limited to the sub-diaphragmatic region with or without pelvic lymph nodes

   * a. No more than a total of 5 lesions on PSMA PET/CT scan (each lesion defined as positive with standardized uptake value (SUV) > liver uptake and CT scan correlate)
   * b. No disease outside of the pelvic and sub-diaphragmatic para-aortic lymph nodes
   * c. At least one lesion in the sub-diaphragmatic para-aortic lymph nodes
   * d. Non-bulky nodal disease (ie, tumor <5 cm)
4. Prior pelvic radiation with disease response

   * a. Definitive radiation therapy to the prostate with or without treatment of the pelvic lymph nodes and/or
   * b. Salvage or adjuvant radiation therapy to the prostate bed following prostatectomy with or without treatment of the pelvic lymph nodes
5. Hormone-sensitive prostate cancer
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
7. Ability to understand the investigational nature, potential risks and benefits of the research study, and willingness to sign the written informed consent and HIPAA document(s)
8. Willingness to fill out quality of life and psychosocial forms
9. Willingness to participate in our institution's Prostate Cancer Database Protocol (ID# 20090767)

Exclusion Criteria:

1. No pathological diagnosis of prostate adenocarcinoma
2. Patient has more than 5 sites of metastatic disease
3. Patient has history of bone and/or visceral metastasis
4. No evidence of disease in the para-aortic lymph nodes
5. No staging with PSMA PET/CT scan
6. History of prior radiation therapy outside the pelvis for prostate cancer
7. Bulky nodal disease >5 cm in tumor size
8. Androgen deprivation therapy (ADT) or chemotherapy in the three months prior to staging PSMA PET/CT scan (suggesting oligoprogressive disease, rather than true oligorecurrent disease) or at time of study enrollment
9. Suspicious radiologic evidence of disease in the prostate on staging PSMA PET/CT scan without confirmatory negative prostate biopsy
10. Implanted hardware which limits treatment planning or delivery (determined by treating physician)
11. Castration-resistant prostate cancer (history of rising PSA with serum testosterone level <50 ng/dL)
12. Patients with ECOG performance status > 2
13. History of inflammatory bowel disease
14. History of malignancy other than prostate cancer except for non-melanoma skin cancer
15. Patients unable to consent or are prisoners
16. Unwilling to fill out quality of life and psychosocial forms
17. Participants with impaired decision-making capacity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to 2 years
  Progression-free survival (PFS) among participants will be assessed during treatment and clinical follow-up. PFS is defined as the time from start of treatment until any of the following: Biochemical failure, escalation of therapy, radiological evidence of disease progression or death of any cause. Radiological evidence of disease progression will be assessed by the treating physician using the Response Evaluation Criteria in prostate-specific membrane antigen (PSMA) PET/CT (RECIP) version 1.0.

SECONDARY OUTCOMES:
Biochemical Failure-Free Survival (FFS) | Up to 2 years
  Biochemical failure-free survival among participants will be assessed during treatment and clinical follow-up. Biochemical failure-free survival is defined as the time from study enrollment to time of biochemical failure. Biochemical failure, as adapted from the Prostate Cancer Working Group 2 (PCWG2), is defined as when prostate-specific antigen (PSA) level increases ≥ 25% and ≥ 2 ng/mL above the nadir, which is confirmed by a second value obtained three or more weeks later.
Metastasis-Free Survival | Up to 2 years
  Metastasis-free survival among participants will be assessed during treatment and clinical follow-up. Metastasis-free survival is defined as the time from study enrollment to clinical or radiological evidence of metastatic disease or death.
Overall Survival (OS) | Up to 2 years
  Overall survival (OS) among participants will be assessed. OS is defined as the time from study enrollment to death of any cause.
Median Cause Specific Survival | Up to 2 years
  Median case specific survival among participants will be assessed. Median cause specific survival is defined as the time from study enrollment to death secondary to prostate cancer.
Proportion of Participants Undergoing Escalation of Therapy | Up to 2 years
  The proportion of participants undergoing escalation of therapy will be reported. Escalation of therapy is defined as subsequent course of radiation therapy or change in systemic therapy (except for intolerable side effects).
Proportion of Participants Experiencing Cumulative Late Grade ≥ 2 Treatment-Related Toxicity | Up to 2 years
  The proportion of participants experience late grade ≥ 2 treatment related toxicity between 90 days and two years following para-aortic radiation therapy (PA-RT) will be reported. Late toxicity is defined as Grade ≥ 2 treatment-related toxicities occurring more than 90 days after completing para-aortic radiation therapy (PA-RT). The severity of the reactions to the treatment will be assessed according to using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Change in Quality of Life Scores: EPIC 26 Short Form | Up to 2 years
  Health-related Quality of Life (HRQOL) will be measured using the Expanded Prostate Cancer Index Composite 26 Short Form (EPIC-26) to evaluate patient function and satisfaction after prostate cancer treatment. EPIC-26 is a short form version of the Expanded Prostate Cancer Index Composite, and is a validated comprehensive instrument developed to measure the health-related quality of life among men with prostate cancer. EPIC-26 consists of 26 items under 5 domains of urinary incontinence, urinary irritative/obstructive, bowel, sexual, and hormonal. Response options for each item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
Change in Quality of Life Scores: HADS | Up to 2 years
  Health-related Quality of Life (HRQOL) will be measured using the Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS is a validated instrument used to measure patient symptoms of anxiety and depression. The HADS questionnaire consists of six questions, three questions each in two domains, HADS-Anxiety and HADS-Depression. Scores in each domain range from 0-9, with higher scores representing greater levels of anxiety and depression.
Change in Quality of Life Scores: IPSS | Up to 2 years
  Health-related quality of life (HRQOL) will be measured using the International Prostate Symptom Score (IPSS) to evaluate patient urinary function and quality of life. There are 7 questions related to urinary function. Responses are on a scale from 0 ("not at all") to 5 ("almost always"), with higher scores indicating higher levels of urinary dysfunction. There is one quality of life question related to urinary symptoms. Responses are on a scale from 0 ("delighted") to 6 ("terrible"). Responses will be tabulated for a composite score.
Complete Early Response Rate | Up to 2 years
  The Complete Early Response rate among participants will be reported. Complete Early Response is defined as seen as on the 3-month post-PA-RT PSMA PET/CT scan using the Response Evaluation Criteria in prostate-specific membrane antigen (PSMA) PET/CT (RECIP) version 1.0; or a PSA level ≤ 0.1 ng/mL. A composite of these two evaluations will be used to determine the complete early response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Rich, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No